CLINICAL TRIAL: NCT01265771
Title: Optimizing Diagnostics And Therapy Of Arrhythmia And Syncope Events Using Intelligent Telemetric Solutions. Diagnostics Of Arrhythmia In Children
Brief Title: Optimizing Diagnostics Of Arrhythmia Events In Children Using Intelligent Telemetric Solutions
Acronym: TELEMARC2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Prof. Lukasz Szumowski MD PhD, Institute of Cardiology, Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UDAPOIG.01.03.01-00-068/09-00B
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Arrhythmia; Children
Keywords: Arrhythmia; Children
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telemetry ordered by a Cardiologist (Experimental)
  Interventions: Device: Prolonged telemetric Full Disclosure ECG recording.
- 24 hours standard Holter monitoring (Experimental)
  Interventions: Device: Repeated 24 hours ECG Holter monitoring
- Telemetry ordered by a Pediatrician (Experimental)
  Interventions: Device: Prolonged telemetric Full Disclosure ECG recording.

INTERVENTIONS:
Device: Prolonged telemetric Full Disclosure ECG recording. — Thirty days Telemetric Full Disclosure ECG monitoring; subsequently analyzed in the Event Holter monitoring mode
  Other Names: Pocket ECG, Medicalgorithmics
  Arms: Telemetry ordered by a Cardiologist; Telemetry ordered by a Pediatrician
Device: Repeated 24 hours ECG Holter monitoring — Repeated 24 hours ECG Holter monitoring
  Arms: 24 hours standard Holter monitoring

SUMMARY:
The purpose of this study is to assess efficacy of prolonged Full Disclosure electrocardiogram (ECG) monitoring and signal analysis using advanced telemetric technology to diagnose arrhythmia in comparison with standard diagnostic procedure.

DETAILED DESCRIPTION:
Irregular and/or rapid beating of the heart called heart palpitations can occur in individuals without heart disease and the reasons for their palpitations are unknown. Together with heart palpitations silent arrhythmia may be present that could lead to serious complications (eg. stroke). In others, palpitations result from heart rhythm disturbances, sometimes life threatening. Standard diagnostic methods such as 24 hours Holter electrocardiogram (ECG) monitoring or Event Holter do not guarantee early diagnosis of the arrhythmia. Prolonged heart rhythm recording and analysis using an automatic full disclosure telemetric device can increase probability of arrhythmia diagnosis and early administration of applicable treatment. Study patients will be diagnosed using standard Holter ECG monitoring, Event Holter or 30 days telemetric ECG monitoring. Efficacy of telemetric monitoring in diagnosis of cardiac arrhythmia will be assessed in comparison with the standard Holter monitoring and Event Holter

ELIGIBILITY:
Inclusion Criteria:

* History of symptoms that can be potentially caused by cardiac arrhythmia occuring at least 4 times a year
* Ability to operate the telemetric device at home
* Informed consent undersigned by the parents
* Informed consent undersigned by the child if over 16 years of age

Exclusion Criteria:

* Previously recorded tachycardia evidence
* Wolff Parkinson White syndrome
* Inability to operate the telemetric device at home
* Inability to comply with the study protocol

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Recording of symptomatic or life threatening arrhythmia event | within 30 days since the start of monitoring
  ECG monitoring is conducted until occurrence of symptomatic arrhythmia or life threatening arrhythmia but not longer than 30 days. Patients in the control group will have standard ECG Holter monitoring repeated twice

SECONDARY OUTCOMES:
Occurrence of silent (asymptomatic) arrhythmia event | within 30 days since the start of monitoring
Verification of patient self assessment based on the Quality of Life questionnaire and European Heart Rhythm Association (EHRA) scale against evidence of cardiac arrhythmia occurrence | within 30 days since the start of monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szumowski, Prof. MD PhD, Study Chair — National Institute of Cardiology, Warsaw, Poland; Katarzyna Bieganowska, Prof. MD PhD, Principal Investigator — Children's Memorial Health Institute
Locations (3):
- Poland (3):
  - Medical University of Warsaw Department of Pediatric Cardiology and General Pediatrics, Warsaw
  - Institute of Cardiology, Warsaw
  - The Children's Memmorial Health Institute, Warsaw